CLINICAL TRIAL: NCT03594851
Title: Evaluation of the Benefits of Individualized Advice Administration on Quality of Sleep for the Elderly Living at Home Prospective, Monocentric and Open Study
Brief Title: Evaluation of the Benefits of Individualized Advice Administration on Quality of Sleep for the Elderly Living at Home
Acronym: CISPAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier de la Region de Mulhouse et Sud Alsace (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GHR 924; ID RCB 2017-A02815-48 (Registry Identifier: Agence Nationale de Sécurité du Médicament et des Produits de Santé)
Record Dates: First submitted 2018-05-22; First posted 2018-07-20 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2018-07

CONDITIONS: Sleep Disorder; Complaint, Subjective Health
Keywords: quality of sleep; elderly; health education; quantity of sleep; caregiver's burden
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders; Health Education | interventions — Activities of Daily Living; Mental Status and Dementia Tests; Quality of Life; Amyloid beta-Protein Precursor

STUDY DESIGN:
Intervention Model Description: Administration of individualized advice to older people living at home complaining of sleep disorders
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Administration of individualized advice (Experimental): Administration of individualized advice to improve the quality of older people's sleep, based on the following interventions :
  Pittsburgh Sleep Quality Index, Sleep diary, Mini Mental State Examination, Autonomy assessment (Katz Index of Independence in Activities of Daily Living
  & Lawton Instrumental Activities of Daily Living), Neuropsychiatric Inventory (Cummings) for the caregiver, if applicable, Mini Zarit Caregiver Burden Scale, for the caregiver, if applicable, Cornell Scale for Depression in Dementia, Quality of Life in Alzheimer's Disease, Neuropsychiatric Inventory
  Interventions: Behavioral: Pittsburgh Sleep Quality Index; Behavioral: Sleep diary; Behavioral: Katz Index of Independence in Activities of Daily Living; Behavioral: Lawton Instrumental Activities of Daily Living; Behavioral: Neuropsychiatric Inventory (Cummings); Behavioral: Mini Zarit Caregiver Burden Scale, for the caregiver; Behavioral: Mini Mental state examination; Behavioral: Cornell Scale for Depression in Dementia; Behavioral: Quality of Life in Alzheimer's Disease

INTERVENTIONS:
Behavioral: Pittsburgh Sleep Quality Index — The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score, and takes 5-10 minutes to complete. Developed by researchers at the University of Pittsburgh, the PSQI is intended to be a standardized sleep questionnaire for clinicians and researchers to use with ease and is used for multiple populations. The questionnaire has been used in many settings, including research and clinical activities, and has been used in the diagnosis of sleep disorders. Clinical studies have found the PSQI to be reliable and valid in the assessment of sleep problems to some degree, but more so with self-reported sleep problems and depression-related symptoms than actigraphic measures.
  Other Names: PSQI
Behavioral: Sleep diary — A sleep diary is a record of a patient's sleep patterns and habits that can be extremely useful in helping doctors make a diagnosis of a sleep disorder and better determine if a sleep study should be prescribed.
Behavioral: Katz Index of Independence in Activities of Daily Living — Katz Activities of Daily Living is a validated tool to assess functional status as a measurement of the elder's ability to perform activities of daily living independently. Elders are scored yes/no for independence in each of six functions. A score of 6 indicates full function, 4 indicates moderate impairment, and 2 or less implies severe functional impairment.
  Other Names: Katz ADL
Behavioral: Lawton Instrumental Activities of Daily Living — Lawton's Instrumental Activities of Daily Living (IADL) scale was developed to assess more complex activities (termed "instrumental activities of daily living") necessary for functioning in community settings (e.g., shopping, cooking, managing finances). The capacity to handle these complex functions normally is lost before basic "activities of daily living" which are measured by Activities of Daily Living scales. Therefore, assessing Instrumental Activities of Daily Living may identify incipient decline in older adults who are otherwise capable and healthy.The Lawton Instrumental Activities of Daily Living scale takes approximately 10 to 15 minutes to administer. It contains 8 items that are rated with a summary score from 0 (low functioning) to 8 (high functioning). This scale can be administered through an interview or by a written questionnaire. The patient or a caregiver who is familiar with the patient can provide the answers.
  Other Names: IADL
Behavioral: Neuropsychiatric Inventory (Cummings) — Neuropsychiatric Inventory is submitted to the caregiver, if the patient has a Mini Mental State Examination score between 10 and 20.
  The Neuropsychiatric Inventory (NPI) was developed by Cummings et al. (1994) to assess dementia-related behavioral symptoms which they felt other measures did not sufficiently address. The NPI originally examined 10 sub-domains of behavioral functioning: delusions, hallucinations, agitation/aggression, dysphoria, anxiety, euphoria, apathy, disinhibition, irritability/lability, and aberrant motor activity. Two more sub-domains have been added since its development: night-time behavioral disturbances and appetite and eating abnormalities (Cummings, 1997). This wide variety of domains means that, unlike other dementia measures, the NPI is able to screen for multiple types of dementia, not just Alzheimer's Disease.
  Other Names: NPI
Behavioral: Mini Zarit Caregiver Burden Scale, for the caregiver — Mini Zarit Caregiver Burden Scale, for the caregiver, if the patient has a Mini Mental State Examination score between 10 and 20.
Behavioral: Mini Mental state examination — It is an 11-question tool to evaluate cognitive functions. The maximum score is 30. A score of 23 or lower is indicative of cognitive impairment. The Mini Mental state examination takes only 5-10 minutes to administer and is therefore practical to use repeatedly and routinely.
  The MMSE has been validated and extensively used in both clinical practice and research, since its creation in 1975
  Other Names: MMSE
Behavioral: Cornell Scale for Depression in Dementia — The Cornell scale For Depression in Dementia is a scoring system specifically developed to assess signs and symptoms of major depression in patients with dementia. The 19 parameters measured are clustered into five groups: mood-related signs, behavioural disturbances, physical signs, cyclic functions and ideational disturbances. The Cornell scale For Depression in Dementia has been shown to be sensitive, reliable and valid for assessing depression in patients with Alzheimer's disease.
Behavioral: Quality of Life in Alzheimer's Disease — The Quality of Life in Alzheimer's Disease is a brief, 13-item measure designed specifically to obtain a rating of the patient's Quality of Life from both the patient and the caregiver. It was developed for individuals with dementia, based on patient, caregiver, and expert input, to maximize construct validity, and to ensure that the measure focuses on quality of life domains thought to be important in cognitively impaired older adults. It uses simple and straightforward language and responses & includes assessments of the individual's relationships with friends and family, concerns about finances, physical condition, mood, and an overall assessment of life quality
  Other Names: QOL-AD

SUMMARY:
Sleep disorder is often a complaint from the older people. Prevalence of sleep disorder increases with aging and reaches between 20 to 45% of the people of 65 years old and more. Sleep physiologically changes with aging. Sleep can also be disturbed by other factors such as intercurrent or related chronic pathologies, environmental change (institutionalized, death of a spouse…), or some medical treatments. Regardless of interindividual variabilities, normative criteria have been defined by a meta-analysis: insomnia can be diagnosed if night wakings are more than 60min and/or if sleep latency is more than 30 minutes.

Various studies have proved the major role of sleep on health and wellbeing. Sleep disorders have an impact on the quality of perception of health and on the quality of life of people and their spouse. According to the French High Health Authority recommendations, sleep diary and validated scales are the tools to use to investigate sleep disorders.

Results from previous studies brought us to consider sleep complaint more specifically and adjust to the heterogeneous population of the investigator's hospital with a subjective approach. This work intends to offer a program of individualized advice to older patients with no cognitive impairment, or with a mild or moderate cognitive impairment, who complain about their sleep quality. Patients with a moderate cognitive impairment who have a caregiver at home can also join the study. The main objective of the study is to evaluate the impact of individualized care for sleep disorders on quality of sleep using the Pittsburgh Sleep Quality Index which validity was demonstrated among the elderly.

ELIGIBILITY:
Inclusion Criteria:

1. Patient giving a signed informed consent
2. Patient complaining about their sleep
3. Patient living at home
4. Patient with a Mini Mental State Examination score of 10 or more If the Mini Mental State Examination score is between 10 and 20, caregiver living at home able and willing to be in charge of a sleep calendar
5. Patient able to fill in questionnaires

Exclusion Criteria:

1. Patient living in a senior living facility
2. Patient legally protected
3. Patient with a psychotic decompensation
4. Patient with a sleep pathology
5. Patient with a Lewy body disease at the time of enrollment
6. Patient with no health insurance

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2019-07-08 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of the benefits of individualized advice administration on sleep quality for the elderly living at home and complaining about their sleep | Through study completion, an average of 6 months
  Evolution of the Pittsburgh Sleep Quality Index. The global PSQI score is calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.

SECONDARY OUTCOMES:
Impact of a specific follow-up on quantity of sleep of elderly complaining about their sleep | Through study completion, an average of 6 months
  Review of the sleep diaries to evaluate the impact on the quantity of sleep
Impact of a specific follow up on quality of life of elderly complaining about their sleep | Through study completion, an average of 6 months
  Evolution of the Mini Mental state examination score : Any score greater than or equal to 24 points (out of 30) indicates a normal cognition. Below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment
Impact of a specific follow up on quality of life of elderly complaining about their sleep | Through study completion, an average of 6 months
  Evolution of the frequency of the patient's falls
Impact of a specific follow up on quality of life of elderly complaining about their sleep | Through study completion, an average of 6 months
  Evolution of the Cornell Scale for Depression in Dementia score : The interviews focus on depressive symptoms and signs occurring during the week preceding the interview. Each item is rated for severity on a scale of 0-2 (0=absent, 1=mild or intermittent, 2=severe). The item scores are added. Scores above 10 indicate a probable major depression; scores above 18 indicate a definite major depression; scores below 6 as a rule are associated with absence of significant depressive symptoms.
Impact of a specific follow up on quality of life of elderly complaining about their sleep | Through study completion, an average of 6 months
  Evolution of the Quality of Life in Alzheimer's Disease questionnaire score : The Quality Of Life - Alzheimer Disease questionnaire is a brief, 13-item measure designed specifically to obtain a rating of the patient's Quality of Life from both the patient and the caregiver. Caregivers complete the measure as a questionnaire about their patients' Quality Of Life, while patients complete it in interview format about their own Quality Of Life. The measure consists of 13 items, rated on a four point scale, with 1 being poor and 4 being excellent. Total scores range from 13 to 52.
Impact of a specific follow up on quality of life of elderly complaining about their sleep | Through study completion, an average of 6 months
  Evolution of the Instrumental Activities of Daily Living questionnaire scores : The Lawton Instrumental Activities of Daily Living scale takes approximately 10 to 15 minutes to administer. It contains 8 items that are rated with a summary score from 0 (low functioning) to 8 (high functioning). This scale can be administered through an interview or by a written questionnaire. The patient or a caregiver who is familiar with the patient can provide the answers.
Impact of a specific follow up on quality of life of elderly complaining about their sleep | Through study completion, an average of 6 months
  Evolution of the Katz Activities of Daily Living scores : Elders are scored yes/no for independence in each of six functions. A score of 6 indicates full function, 4 indicates moderate impairment, and 2 or less implies severe functional impairment.
Impact of a specific follow up on quality of life of elderly complaining about their sleep | Through study completion, an average of 6 months
  Evolution of the Neuropsychiatric Inventory score. The Neuropsychiatric Inventory uses a structured, caregiver-based interview format to assess 10 behavioral domains (Delusions, Hallucinations, Agitation, Dysphoria, Anxiety, Apathy, Irritability, Euphoria, Disinhibition, and Aberrant motor behavior). Two additional domains (Nighttime behavioral disturbance, and Appetite/weight changes) are often added. The presence of problematic behaviors in each domain is assessed by asking an informant a screening question followed by a series of yes/no questions. The caregiver or surrogate reporter is then asked to rate the frequency of occurrence of that domain of behaviors. The same behaviors are then rated on level of severity (1 = mild, 2 = moderate, 3 = severe). The domain total score is the product of the frequency score multiplied by the severity score for that behavioral domain. A Neuropsychiatric Inventory total score is obtained by summing all the individual domain total scores.
Impact of a specific follow up on quality of life of elderly complaining about their sleep | Through study completion, an average of 6 months
  Evolution of the psychotropic drug consumption (how many and which type)
Impact of a specific follow up on quality of life of caregivers of elderly complaining about their sleep | Through study completion, an average of 6 months
  Evolution of the Quality of Life in Alzheimer's Disease questionnaire score : The QOL-AD is a brief, 13-item measure designed specifically to obtain a rating of the patient's Quality of Life from both the patient and the caregiver. Caregivers complete the measure as a questionnaire about their patients' Quality Of Life, while patients complete it in interview format about their own Quality Of Life. The measure consists of 13 items, rated on a four point scale, with 1 being poor and 4 being excellent. Total scores range from 13 to 52.
Impact of a specific follow up on the burden of caregivers of elderly complaining about their sleep | Through study completion, an average of 6 months
  Evolution of the 7 item Zarit Care Burden Interview scale score. Points are assigned to each items as follows : never=0; sometimes=0,5 ; often=1 Total score is the sum of all items, 0-2 : Little or no burden 2-3,5: Mild to moderate burden 3,5-5,5: Moderate to severe burden 5,5-7: Severe burden

CONTACTS AND LOCATIONS:
Overall Officials: Anna Derajinski, MD, Principal Investigator — Groupe Hospitalier de la Region de Mulhouse et Sud Alsace
Locations (1):
- GHRMSA, Mulhouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ohayon MM, Lemoine P. [Sleep and insomnia markers in the general population]. Encephale. 2004 Mar-Apr;30(2):135-40. doi: 10.1016/s0013-7006(04)95423-1. French. PMID 15107715
- [Background] Kamel NS, Gammack JK. Insomnia in the elderly: cause, approach, and treatment. Am J Med. 2006 Jun;119(6):463-9. doi: 10.1016/j.amjmed.2005.10.051. PMID 16750956
- [Background] Corman B, Leger D. [Sleep disorders in elderly]. Rev Prat. 2004 Jun 30;54(12):1281-5. French. PMID 15461045
- [Background] Edinger JD, Bonnet MH, Bootzin RR, Doghramji K, Dorsey CM, Espie CA, Jamieson AO, McCall WV, Morin CM, Stepanski EJ; American Academy of Sleep Medicine Work Group. Derivation of research diagnostic criteria for insomnia: report of an American Academy of Sleep Medicine Work Group. Sleep. 2004 Dec 15;27(8):1567-96. doi: 10.1093/sleep/27.8.1567. PMID 15683149
- [Background] Silva J, Truzzi A, Schaustz F, Barros R, Santos M, Laks J. Impact of insomnia on self-perceived health in the elderly. Arq Neuropsiquiatr. 2017 May;75(5):277-281. doi: 10.1590/0004-282X20170031. PMID 28591386
- [Background] Nguyen-Michel VH, Vecchierini MF. Exploration of sleep disorders in the elderly: which particularities? Geriatr Psychol Neuropsychiatr Vieil. 2016 Dec 1;14(4):429-437. doi: 10.1684/pnv.2016.0634. PMID 27976622
- [Background] Vecchierini MF. [Sleep disturbances in Alzheimer's disease and other dementias]. Psychol Neuropsychiatr Vieil. 2010 Mar;8(1):15-23. doi: 10.1684/pnv.2010.0203. French. PMID 20215095
- [Background] McKeith IG, Boeve BF, Dickson DW, Halliday G, Taylor JP, Weintraub D, Aarsland D, Galvin J, Attems J, Ballard CG, Bayston A, Beach TG, Blanc F, Bohnen N, Bonanni L, Bras J, Brundin P, Burn D, Chen-Plotkin A, Duda JE, El-Agnaf O, Feldman H, Ferman TJ, Ffytche D, Fujishiro H, Galasko D, Goldman JG, Gomperts SN, Graff-Radford NR, Honig LS, Iranzo A, Kantarci K, Kaufer D, Kukull W, Lee VMY, Leverenz JB, Lewis S, Lippa C, Lunde A, Masellis M, Masliah E, McLean P, Mollenhauer B, Montine TJ, Moreno E, Mori E, Murray M, O'Brien JT, Orimo S, Postuma RB, Ramaswamy S, Ross OA, Salmon DP, Singleton A, Taylor A, Thomas A, Tiraboschi P, Toledo JB, Trojanowski JQ, Tsuang D, Walker Z, Yamada M, Kosaka K. Diagnosis and management of dementia with Lewy bodies: Fourth consensus report of the DLB Consortium. Neurology. 2017 Jul 4;89(1):88-100. doi: 10.1212/WNL.0000000000004058. Epub 2017 Jun 7. PMID 28592453
- [Background] McCurry SM, Logsdon RG, Teri L, Vitiello MV. Sleep disturbances in caregivers of persons with dementia: contributing factors and treatment implications. Sleep Med Rev. 2007 Apr;11(2):143-53. doi: 10.1016/j.smrv.2006.09.002. Epub 2007 Feb 6. PMID 17287134
- [Background] Thomas P, Hazif-Thomas C, Pareault M, Vieban F, Clement JP. [Sleep disturbances in home caregivers of persons with dementia]. Encephale. 2010 Apr;36(2):159-65. doi: 10.1016/j.encep.2009.06.010. Epub 2009 Sep 23. French. PMID 20434634
- [Background] Gauriau C, Raffray T, Choudat D, Corman B, Leger D. [Objective improvement of sleep disorders in the elderly by a health education program]. Presse Med. 2007 Dec;36(12 Pt 1):1721-31. doi: 10.1016/j.lpm.2007.07.002. Epub 2007 Jul 30. French. PMID 17659860
- [Background] Crawford-Achour E, Castro-Lionard K, Tardy M, Trombert-Paviot B, Barthelemy JC, Gonthier R. [Successful aging: how to improve its occurrence in the elderly?]. Geriatr Psychol Neuropsychiatr Vieil. 2012 Jun;10(2):207-14. doi: 10.1684/pnv.2012.0318. French. PMID 22713850
- [Background] E. Crawford-Achour et al. Can subjective sleep quality, evaluated at the age of 73, have an influence on successful aging? The PROOF study. Open Journal of Preventive Medicine 4 (2014) 51-56. http://dx.doi.org/10.4236/ojpm.2014.42008
- [Background] Grandner MA, Kripke DF, Yoon IY, Youngstedt SD. Criterion validity of the Pittsburgh Sleep Quality Index: Investigation in a non-clinical sample. Sleep Biol Rhythms. 2006 Jun;4(2):129-139. doi: 10.1111/j.1479-8425.2006.00207.x. Epub 2006 Jun 9. PMID 22822303
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Cole JC, Motivala SJ, Buysse DJ, Oxman MN, Levin MJ, Irwin MR. Validation of a 3-factor scoring model for the Pittsburgh sleep quality index in older adults. Sleep. 2006 Jan;29(1):112-6. doi: 10.1093/sleep/29.1.112. PMID 16453989
- [Background] Derouesne C, Poitreneau J, Hugonot L, Kalafat M, Dubois B, Laurent B. [Mini-Mental State Examination:a useful method for the evaluation of the cognitive status of patients by the clinician. Consensual French version]. Presse Med. 1999 Jun 12;28(21):1141-8. French. PMID 10399508
- [Background] Alexopoulos GS, Abrams RC, Young RC, Shamoian CA. Cornell Scale for Depression in Dementia. Biol Psychiatry. 1988 Feb 1;23(3):271-84. doi: 10.1016/0006-3223(88)90038-8. PMID 3337862
- [Background] Novella JL, Dhaussy G, Wolak A, Morrone I, Drame M, Blanchard F, Jolly D. [Quality of life in dementia: state of the knowledge]. Geriatr Psychol Neuropsychiatr Vieil. 2012 Dec;10(4):365-72. doi: 10.1684/pnv.2012.0375. French. PMID 23250016
- [Background] Carney CE, Buysse DJ, Ancoli-Israel S, Edinger JD, Krystal AD, Lichstein KL, Morin CM. The consensus sleep diary: standardizing prospective sleep self-monitoring. Sleep. 2012 Feb 1;35(2):287-302. doi: 10.5665/sleep.1642. PMID 22294820
- [Background] French High Health Authority. Alzheimer Disease and related pathologies : medical follow up of the natural caregivers. Guidelines (french recommendations) https://www.has-sante.fr/portail/upload/docs/application/pdf/2010-03/maladie_dalzheimer_-_suivi_medical_des_aidants_naturels_-_argumentaire_2010-03-31_15-38-54_749.pdf
- [Background] Higginson IJ, Gao W, Jackson D, Murray J, Harding R. Short-form Zarit Caregiver Burden Interviews were valid in advanced conditions. J Clin Epidemiol. 2010 May;63(5):535-42. doi: 10.1016/j.jclinepi.2009.06.014. PMID 19836205
- [Background] Bedard M, Molloy DW, Squire L, Dubois S, Lever JA, O'Donnell M. The Zarit Burden Interview: a new short version and screening version. Gerontologist. 2001 Oct;41(5):652-7. doi: 10.1093/geront/41.5.652. PMID 11574710